CLINICAL TRIAL: NCT03056742
Title: A Single Arm, Open Label, Multicentric, Clinical Study Assessing the Efficacy and Safety of Stempeucel® (ex Vivo Cultured Adult Bone Marrow Derived Allogeneic Mesenchymal Stem Cells) in Patients With CLI Due to Buerger's Disease
Brief Title: A Clinical Trial to Study the Efficacy and Safety of Stempeucel® in Patients With CLI Due to Buergers Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Form 46 from DCGI for the manufacturing & commercial marketing of Stempeucel® directs Stempeutics to conduct PMS study. Hence this study is being terminated.
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRPL/CLI/10-11/001 Version 4
Record Dates: First submitted 2017-01-23; First posted 2017-02-17 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Critical Limb Ischemia Due to Buerger's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cells (Experimental): Patients will receive intramuscular and local injection of stempeucel(R) in addition to standard protocol of care
  Interventions: Biological: Stempeucel(R)

INTERVENTIONS:
Biological: Stempeucel(R) — Ex vivo cultured adult bone marrow derived allogeneic mesenchymal stem cells

SUMMARY:
This study is being conducted as an extension of the phase II clinical trial SRPL/CLI/10-11/001 (NCT01484574). The CDSCO has recommended flexibility for continued clinical study in consultation with ICMR, as per recommendation of Cellular biology based therapeutic drug evaluation committee (CBBTDEC).

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of intramuscular injection of stempeucel(R) (Ex vivo cultured adult bone marrow derived allogeneic mesenchymal stem cells) in Critical Limb Ischemia due to Buerger's Disease

ELIGIBILITY:
Inclusion Criteria:

1. Buerger's disease as diagnosed by Shionoya criteria
2. Males or females (willing to use accepted methods of contraception during the course of the study) in the age group of 18-65 yrs.
3. Established CLI in the study limb, clinically and hemodynamically confirmed as per Rutherford- III-5;
4. Patients in Rutherford- III-6 if gangrene extending maximally up to the head of metatarsal but limited to toes (patients with wet gangrene must undergo wound debridement / amputation before screening) .
5. Patients having infrapopliteal occlusive disease with rest pain and ischemic ulcer/necrosis (patients should have at least one measureable ulcer), who are not eligible for or have failed traditional revascularization treatment as per the investigators judgment (No option patients) .
6. ABPI ≤ 0.6 or ankle pressure ≤ 50 mm Hg.
7. Patients who are able to understand the requirements of the study, and willing to provide voluntary written informed consent and video consent, abide by the study requirements, and agree to return for required follow-up visits.

Exclusion Criteria:

1. Patients with CLI indicated for major amputation during screening
2. Atherosclerotic PAD
3. Ulcers with exposure of tendon and/bone in the shin region.
4. Previous above trans metatarsal amputation in study limb
5. Any Lumbar sympathectomy procedure performed less than 90 days prior to the screening
6. Patients with gait disturbance for reasons other than CLI
7. Diagnosis of diabetes mellitus (type 1 or type 2)
8. Patients having left ventricular ejection fraction < 35%
9. Patients suffering from clinically relevant peripheral neuropathy
10. History of stroke or myocardial infarction
11. Patients who are contraindicated for MRA
12. Patients with DVT in any limb.
13. Patients who have clinically serious and/or unstable inter-current infection, medical illnesses or conditions that are uncontrolled or whose control, in the opinion of the Investigator, may be jeopardized by participation in this study or by the complications of this therapy
14. Documented terminal illness or cancer or any concomitant disease process with a life expectancy of <1 year
15. Patients already enrolled in another investigational drug trial or completed within 3 months or those who have received stem cells in the past
16. Patient with known hypersensitivity to the constituents of the stempeucel®- dimethyl sulfoxide (DMSO) or human serum albumin (HSA)
17. History of severe alcohol or drug abuse within 3 months of screening
18. Hb% < 10 gm% for males, Hb% < 9 gm% for females, serum creatinine ≥ 2mg%, serum Total Bilirubin ≥2mg%
19. Pregnant and lactating women
20. Patients tested positive for HIV 1 & 2, HCV, HBV, CMV, RPR antibodies and for HBsAg antigen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-20 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Relief of the rest pain | 6 months
Reduction of ulcer area in the target limb | 6 months

SECONDARY OUTCOMES:
Total walking distance | 6 months and 24 months
Major amputation free survival | 6 months and 24 months
Ankle brachial pressure index (ABPI) - measured by Doppler | 6 months and 24 months
Quality of life (QOL) by King's College VascuQOL questionnaire | 6 months and 24 months
Angiogenesis - collateral blood vessels by Magnetic resonance angiogram (MRA) | 6 months and 24 months

OTHER OUTCOMES:
The type of adverse events AE(s), number of AE(s) and proportion of patients with AE(s). | 6 months and 24 months
CVS mortality | 6 months and 24 months
All-cause mortality | 6 months and 24 months

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Department of Vascular and Endovascular Surgery, M. S. Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Department of Surgical Disciplines, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Department of Vascular Surgery, Madras Medical College, Chennai, Tamil Nadu
  - Department of Vascular Surgery, Sri Ramchandra Medical College, Chennai, Tamil Nadu
  - Saveetha Medical College & Hospital, Chennai, Tamil Nadu
  - SRM Medical College Hospital and Research Centre, Chennai, Tamil Nadu
  - Health Point Hospital, Kolkata, West Bengal
  - Nightingale Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No